CLINICAL TRIAL: NCT05433610
Title: Is Non-invasive Ventilation Effective in Improving the Exercise Capacity in Patients With Cardiac Heart Failure?: A Randomized Controlled Trial
Brief Title: Non-invasive Ventilation in Patients With Cardiac Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Guillermo A. Mazzucco, Principal Investigator, University of Gran Rosario
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 344/2021
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure
Keywords: Rehabilitation; Exercise Test; Heart Failure; Aerobic Exercise
MeSH Terms: conditions — Heart Failure | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Interventional, crossover, randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Constant Treadmill Load Test (CTLT) using non-invasive ventilation (NIV) (Experimental): Exercise capacity testing using PS in HF patients
  Interventions: Device: Non-invasive Ventilation
- Constant Treadmill Load Test (CTLT) using NIV (Experimental): Exercise capacity testing using CPAP in HF patients
  Interventions: Device: Non-invasive Ventilation
- Constant Treadmill Load Test (CTLT) without NIV (Active Comparator): Exercise capacity testing without NIV in HF patients
  Interventions: Device: Non-invasive Ventilation

INTERVENTIONS:
Device: Non-invasive Ventilation — Exercise capacity testing using the device
  Other Names: Noninvasive Ventilations

SUMMARY:
Patients with heart failure (HF) have a reduced exercise tolerance as the main result of the disease. This exercise intolerance is due to heart conditions, but also to dysfunction of the respiratory and peripheral muscles. Various factors such as chronic hypoxia, oxidative stress, nutritional depletion, peripheral muscle disuse, effects of medications, and sympathetic-vagal imbalance are major contributors to deconditioning. In this scenario, the use of non-invasive ventilatory support (NIV) arises as an adjunct to cardiac rehabilitation in the attempt to improve the functional capacity of patients, since NIV reduces work of breathing, improves oxygenation and increases lung compliance associated with improved ejection volume, due to increased intrathoracic pressure.

DETAILED DESCRIPTION:
The main objective is to evaluate whether the use of NIV during Constant Treadmill Load Tests (CTLT) enhances exercise performance in Cardiac Heart Failure (CHF) patients on a treadmill.

Each recruited patient will be evaluated on 4 occasions, with two different evaluations, an incremental test (IT) to find out the maximum aerobic speed reached and then, in randomized order, three CTLT at 85% of the maximum reached in the IT . Two of the three CTLT will be performed with the use of NIV, with PS (IPAP 10cmH2O and EPAP 5cmH2O) and CPAP (5cmH2O) mode, and the rest will be without the use of NIV. The main study variable will be the time tolerated on the treadmill during CTLT.

Participants will have 5 minutes to adapt to NIV, 5-minute warm-up at 50% and then will start with the CTLT at 85% of the maximum aerobic speed reached in the IT.

In total, each patient will be evaluated four times on four different visits.

Sample size: For the sample's calculation, the maximum time in CTLC was chosen as the main study variable because it is a sensitive measure to detect changes after interventions (both pharmacological and non-pharmacological) and widely used in clinical trials. A minimum difference to detect of 100 seconds from previous literature was determined. Taking this data into account, and using a level of α of 0.05, a 1-β power of 0.80, and an effect size of 0.8, the sample size calculation for a paired t-test investigators found that at least 12 participants are needed. The calculation was made using the Gpower 3.1.9.7 software.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction demonstrated by echocardiography ≤ 40% (in the last 12 months).
* NYHA functional class I - III.
* Clinical stability, defined as four weeks prior to the start of the study without hospitalizations.
* Signed informed consent.
* ≥ 18 years of age.

Exclusion Criteria:

* Chronic obstructive pulmonary disease (COPD), unstable angina or significant arrhythmias.
* Myocardial infarction in the last 3 months, primary valve disease and anemia (hemoglobin under 13 g/dl for men or 12 g/dl for women).
* Patients who are smokers or ex-smokers of less than one year.
* Patients with cognitive impairment that prevents the correct understanding of the evaluations.
* Any neuromuscular or osteoarticular condition that limits test performance.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in exercise tolerance | At the end of exercise
  Change in Maximun Walking time tolerated in a Constant Treadmill Load Test (CTLT) in seconds on treadmill between PS, CPAP and WNIT

SECONDARY OUTCOMES:
Change in Dyspnea | At the end of exercise
  Degree of dyspnea will be determined by this validated scale with a result between 0 and 10 points.0: Not at all 0.5: Very, very light (hardly noticeable) 1: Very light, 2: Light, 3: Moderate , 4: Somewhat intense, 5: Intense, 6: Between 5 and 7, 7: Very intense, 8: Between 7 and 9, 9: Very, very intense (almost maximum ), 10: Maximum.
Change in Cardiac Rate | At the end of exercise
  Difference in Cardiac Rate (beats per minute) using a pulse oximetry (Masimo Radical 7) and a heart rate monitor (Polar FT1) between PS, CPAP and WNIT
Change in Oxygen Saturation | At the end of exercise
  Change in Oxygen Saturation using a pulse oximetry (Masimo Radical 7) between PS, CPAP and WNIT
Change in Global Comfort | At the end of exercise
  Change in global comfort according to the device used with Visual Analogue Scale (VAS). The VAS is a 10 cm line with anchor statements on the left (very unpleasant) and on the right (very pleasant) 0-10cm.
Change in Lower Limbs Fatigue | At the end of exercise
  Change in Lower limbs fatigue perception using the Modified Borg Scale (Degree of fatigue will be determined by this validated scale with a result between 0 and 10 points.0: Not at all 0.5: Very, very light (hardly noticeable) 1: Very light, 2: Light, 3: Moderate , 4: Somewhat intense, 5: Intense, 6: Between 5 and 7, 7: Very intense, 8: Between 7 and 9, 9: Very, very intense (almost maximum ), 10: Maximum.
Change in Blood Pressure | At the end of exercise
  Change in Systolic and Dyastolic blood preassure in mmHg at the beginning and at the end.
Change in Recovery heart rate | At the end of exercise
  Change in heart rate (beats per minute) in the first minute, in the second minute and in the third minute after the test, using pulse oximetry (Masimo Radical 7)
Change in the motive for stopping the test | At the end of exercise
  Change in reason for stopping the test. A dichotomous question will be asked regarding the reason for stopping the test, whether it was due to dyspnea or lower limb fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] O'Donnell DE, D'Arsigny C, Raj S, Abdollah H, Webb KA. Ventilatory assistance improves exercise endurance in stable congestive heart failure. Am J Respir Crit Care Med. 1999 Dec;160(6):1804-11. doi: 10.1164/ajrccm.160.6.9808134. PMID 10588589
- [Background] Bittencourt HS, Reis HF, Lima MS, Gomes M Neto. Non-Invasive Ventilation in Patients with Heart Failure: A Systematic Review and Meta-Analysis. Arq Bras Cardiol. 2017 Feb;108(2):161-168. doi: 10.5935/abc.20170001. Epub 2017 Jan 16. PMID 28099587
- [Background] Gosker HR, Wouters EF, van der Vusse GJ, Schols AM. Skeletal muscle dysfunction in chronic obstructive pulmonary disease and chronic heart failure: underlying mechanisms and therapy perspectives. Am J Clin Nutr. 2000 May;71(5):1033-47. doi: 10.1093/ajcn/71.5.1033. PMID 10799364
- [Background] Borghi-Silva A, Carrascosa C, Oliveira CC, Barroco AC, Berton DC, Vilaca D, Lira-Filho EB, Ribeiro D, Nery LE, Neder JA. Effects of respiratory muscle unloading on leg muscle oxygenation and blood volume during high-intensity exercise in chronic heart failure. Am J Physiol Heart Circ Physiol. 2008 Jun;294(6):H2465-72. doi: 10.1152/ajpheart.91520.2007. Epub 2008 Mar 28. PMID 18375714
- [Derived] Mazzucco G, Torres-Castro R, Intelangelo L, Lista-Paz A, Escalante JP, Zumeta-Olaskoaga L, Veiga G, Etxarri AA. Is non-invasive ventilation effective in improving the exercise capacity in patients with cardiac heart failure?: A randomised crossover trial. PLoS One. 2025 Jul 7;20(7):e0327399. doi: 10.1371/journal.pone.0327399. eCollection 2025. PMID 40622949